CLINICAL TRIAL: NCT01856101
Title: A Single Arm, Multicenter, Phase II Study of BEZ235 as Monotherapy in Patients With Locally Advanced or Metastatic Transitional Cell Carcinoma (TCC) After Failure of Platinum Based Chemotherapy.
Brief Title: Study of BEZ235 as Monotherapy in Patients With Transitional Cell Carcinoma After Failure of Platinum Based Chemotherapy
Acronym: BEZ235
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis decided to stop the marketing of BEZ235
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO2012-01; 2012-004123-20 (EudraCT Number); CBEZ235ZBE01T (Other: CB)
Record Dates: First submitted 2012-12-10; First posted 2013-05-17 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma Transitional Cell
Keywords: TCC; Failure of platinum based chemotherapy
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — dactolisib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEZ235, powder (Experimental): * Group 1: patients without PI3K pathway activation; no loss of PTEN and no activating PIK3CA mutation.
  * Group 2: patients with PI3K pathway activation as defined by PIK3CA mutation and/or PTEN loss
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235 — The investigational study drug used in this trial is BEZ235, supplied as 200 mg, 300 mg and 400 mg sachets. BEZ235 is administered continuously twice-daily; complete cycle is 28 days. Starting dose is 300mg PO bid. At cycle 1 day 15, based on a clinical assessment, dose is adjusted for the rest of the study:• If no adverse event (AE) or only mild AE (G1) : the dose will be increase to 400 mg bid• If AE = G2 : the patient will continue at 300 mg bid • If G3 AE or higher : BEZ235 will be interrupt until resolved to ≤ G1 then reduce dose to 200 mg bid
  Other Names: BEZ235 is a potent dual pan class I PI3K and mTOR inhibitor.

SUMMARY:
The mTOR (mammalian Target of Rapamycin) protein is the center of the mTOR pathway that plays an important role in cell growth, proliferation, survival and angiogenesis through sensing and integrating energetic signals from cellular environment. The mTOR protein is composed of two complex, mTOR complex 1 (mTOR C1) and mTOR complex 2 (mTOR C2).

In regards of mTOR pathway dysregulations observed in TCC development, there is a rational to test BEZ23 in advanced TCC. BEZ235 is a pan-class I PI3K inhibitor that, in addition, binds to the catalytic site of mTOR, inhibiting mTOR C1 and mTOR C2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically- or cytologically-confirmed locally advanced or metastatic TCC not amenable to curative surgery or radiation.
2. Documented disease progression (according RECIST 1.1 criteria) after first line platinum-based therapy (given in neoadjuvant/adjuvant or palliative setting).
3. An interval of >4 weeks since last anticancer treatment.
4. Archival paraffin-embedded tumor tissue (block or at least 20 unstained slides) of the primary tumor and/or metastases. The most recent archival tissue is mandatory. Recidive of the disease should lead to perform if possible novel biopsies, as major oncogenic differences are found between primary tumor and secondary lesions.
5. At least one measurable lesion by MRI or CT-scan
6. ECOG performance status 0-1, in stable medical condition
7. Patients must have adequate organ function: Hemoglobin ≥ 9 g/100 ml, neutrophils ≥ 1,000/mm3, platelets ≥ 100,000/mm, INR ≤ 1.5, total serum bilirubin ≤ 1.5 x ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (or <5.0 x ULN if hepatic metastases are present), creatinine £1.5 x ULN, fasting plasma glucose <140mg/dl, HbA1c < 8%.
8. Patients must be over 18 years old and able to give written informed consent.
9. Signed informed consent prior to beginning protocol specific procedure

Exclusion Criteria:

1. Non- TCC bladder cancer
2. More than 2 prior chemotherapy regimens given for palliation.
3. Concurrent malignancy or previous malignancy in the last 3 years prior to start the study treatment (with the exception of a history of adequately treated cervical carcinoma in situ or non-melanoma skin cancer)
4. Patient with active uncontrolled or symptomatic central nervous system (CNS metastases).
5. Significant active cardiac disease including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, or serious cardiac arrhythmias.
6. Other uncontrolled medical condition (active infections requiring antibiotics, bleeding disorders, uncontrolled diabetes …)
7. Other concomitant anticancer therapy.
8. Previous therapy with PI3K and/or mTOR inhibitors (sirolimus, temsirolimus, everolimus)
9. Concomitant drugs such as coumarin and warfarin, and drugs known to induce torsade de pointe, drugs known to be moderate or strong inhibitors or inducers of CYP3A4
10. Pregnancy or risk of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of BEZ235 in patients with palliative TCC | at 16 weeks (radiological evaluation every 8 weeks)
  o Control disease rate at 16 weeks, including complete responses, partial responses and stable diseases according to RECIST criteria.

SECONDARY OUTCOMES:
Determine the safety profile of BEZ235 in patients with advanced TCC | participants will be followed for the duration of hospital stay, an expected average of 16 weeks
  The patient will have an appointment with the investigator on day 15 of cycle 1 and every day 1 of each cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, PhD, Principal Investigator — Centre du Cancer, Cliniques universitaires Saint-Luc
Locations (12):
- Belgium (11):
  - Clinique Saint-Pierre à Ottignies, Ottignies, Brabant Wallon
  - Epicura- RHMS Baudour, Baudour, Hainaut
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Hôpital de Jolimont, Haine-Saint-Paul, Hainaut
  - Centre Hospitalier Wallonie Picarde, Tournai, Hainaut
  - CHU de Liège site du Sart Tilman, Liège, Liège
  - Clinique du Sud Luxembourg, Arlon, Luxembourg
  - CHU de Mont-Godinne, Yvoir, Namur
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique et Maternité Ste Elisabeth, Namur
- Centre Hospitalier de Luxembourg, Luxembourg, Grand-Duché de Luxembourg, Luxembourg